CLINICAL TRIAL: NCT01509937
Title: A Randomized Controlled Trial of Long Term Effect of BCM Guided Fluid Management in MHD Patients
Brief Title: Body Composition Monitor(BCM) Guided Fluid Management in Maintenance Hemodialysis (MHD) Patients
Acronym: BOCOMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Fresenius Medical Care (Shanghai) Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Li Zuo, Clinical professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BOCOMO525
Record Dates: First submitted 2012-01-03; First posted 2012-01-13 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: End Stage Renal Disease
Keywords: end stage renal disease; maintenance hemodialysis; dry weight; bioimpedance spectroscopy analysis; body composition monitor; Fresenius BCM; Ultrafiltration
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BCM Arm (Experimental): BCM measured every 2 months
  Interventions: Device: body bioimpedance spectroscopy device
- Control arm (Sham Comparator): patients care according to standard of care
  Interventions: Device: Device

INTERVENTIONS:
Device: body bioimpedance spectroscopy device — Name of the device is BCM from Fresenius Medical Care D GmbH
  Arms: BCM Arm
Device: Device — participants in control arm will not receive BCM measurement.
  Arms: Control arm

SUMMARY:
It is hypothesized that bioimpedance spectroscope guided fluid management will help patient reach euvolemic status, and increase long term survival.

Background: Bioimpedance analysis (BIA) was helpful in identifying hypervolemia. Observational data using BIA methods showed that hypervolemic patients on maintenance hemodialysis (MHD) suffered from high mortality risk. But it is not clear if BIA guided fluid management can improve MHD patients' survival. The objectives of the BOCOMO study are to evaluate the outcome of BIA guided fluid management comparing with standard care.

Design: This is a multicenter, prospective, randomized, controlled trial. Setting and Participants: More than 1300 participants from 16 clinical sites will be included in the study. The enrollment period will last 6 months, and minimum length of follow-up will not less than 36 months. MHD patients aged more than 18 years but less than 80 years who had been on MHD for at least 3 months and considered suitable candidates will be invited to participate in the study. Participants will be randomized to BIA arm or control arm using 1:1 ratio. A portable whole body bioimpedance spectroscopy device (BCM-Fresenius Medical Care D GmbH) will be used for BIA measurement at baseline for both arm, and every 2 months in BCM arm.

Predictors: BCM guided fluid management and fluid management using standard care.

Outcome and measurements: The primary intent-to-treat analysis compares composite endpoint between BCM arm and control arm. The secondary intent-to-treat analysis compares left ventricular thickness, blood pressure, medication, and incidence and length of hospitalization between BCM arm and control arm. Death, acute myocardial infarction, stroke, peripheral arterial disease will be used as composite endpoint.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of end stage renal disease (ESRD) and need MHD
* age of 18 years or older but 80 years or less
* on MHD for at least 3 months
* dialysis frequency of at least 5 sessions per 2 weeks, not less than 4 hours per session, Kt/V at least 1.2
* urine volume less than 800mL per 24 hours the day before dialysis session,
* bioimpedance analysis not used within recent 3 months
* dry weight regarded as adequate according to the patient's responsible doctor
* the ability to understand and willingness to sign an informed consent statement.

Exclusion Criteria:

* acute infection within 1 month
* active rheumatic disease, or current on cortical steroid medication or cytotoxic medication
* uncontrolled neoplasm
* acute myocardial infarction within 1 month
* congestive heart failure (NYHA 3 - 4)
* stroke within 3 months,
* metallic installation, like contraceptive device, artificial joint(s)
* amputation
* female of childbearing age who has a pregnancy plan, or is pregnant, or on breast feeding
* having a plan to reduce dialysis frequency
* having a renal transplantation plan or planning to transfer to peritoneal dialysis within 3 years
* participating or planning to participate another clinical trial, which will confound the current study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of composite endpoint | during 36 months
  Death, acute myocardial infarction, cerebral thrombosis, cerebral hemorrhage, peripheral arterial disease will be used as composite endpoint.

SECONDARY OUTCOMES:
Change from baseline in Left ventricular thickness once a year | baseline, and once a year during the following 36 months
Change from baseline in Pre-dialysis blood pressure every 2 months | baseline, every 2 months during the following 36 months
Change from baseline in anti-hypertensives DDD every 2 months | Baseline, and every 2 months during the following 36 months
  Defined daily dose (DDD) will be calculated according to WHO recommendation at baseline, and every 2 months thereafter. Trend of DDD change will be compared between the two arms.
Incidence of all cause and congestive heart failure related hospitalization | during the 36 months
  Incidence of all cause and congestive heart failure related hospitalization will be compared between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zuo, MD & PhD, Study Director — Institute of Nephrology, Peking University
Locations (1):
- Institute of Nephrology, Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Wizemann V, Wabel P, Chamney P, Zaluska W, Moissl U, Rode C, Malecka-Masalska T, Marcelli D. The mortality risk of overhydration in haemodialysis patients. Nephrol Dial Transplant. 2009 May;24(5):1574-9. doi: 10.1093/ndt/gfn707. Epub 2009 Jan 7. PMID 19131355
- [Background] Jansen MA, Hart AA, Korevaar JC, Dekker FW, Boeschoten EW, Krediet RT; NECOSAD Study Group. Predictors of the rate of decline of residual renal function in incident dialysis patients. Kidney Int. 2002 Sep;62(3):1046-53. doi: 10.1046/j.1523-1755.2002.00505.x. PMID 12164889
- [Background] Puskar D, Pasini J, Savic I, Bedalov G, Sonicki Z. Survival of primary arteriovenous fistula in 463 patients on chronic hemodialysis. Croat Med J. 2002 Jun;43(3):306-11. PMID 12035137
- [Background] Mizumasa T, Hirakata H, Yoshimitsu T, Hirakata E, Kubo M, Kashiwagi M, Tanaka H, Kanai H, Fujimi S, Iida M. Dialysis-related hypotension as a cause of progressive frontal lobe atrophy in chronic hemodialysis patients: a 3-year prospective study. Nephron Clin Pract. 2004;97(1):c23-30. doi: 10.1159/000077592. PMID 15153764
- [Background] John AS, Tuerff SD, Kerstein MD. Nonocclusive mesenteric infarction in hemodialysis patients. J Am Coll Surg. 2000 Jan;190(1):84-8. doi: 10.1016/s1072-7515(99)00226-4. PMID 10625237
- [Background] Shoji T, Tsubakihara Y, Fujii M, Imai E. Hemodialysis-associated hypotension as an independent risk factor for two-year mortality in hemodialysis patients. Kidney Int. 2004 Sep;66(3):1212-20. doi: 10.1111/j.1523-1755.2004.00812.x. PMID 15327420
- [Background] Tisler A, Akocsi K, Harshegyi I, Varga G, Ferenczi S, Grosz M, Kulcsar I, Locsey L, Samik J, Solt I, Szegedi J, Toth E, Wagner G, Kiss I. Comparison of dialysis and clinical characteristics of patients with frequent and occasional hemodialysis-associated hypotension. Kidney Blood Press Res. 2002;25(2):97-102. doi: 10.1159/000063515. PMID 12077491
- [Background] Pillon L, Piccoli A, Lowrie EG, Lazarus JM, Chertow GM. Vector length as a proxy for the adequacy of ultrafiltration in hemodialysis. Kidney Int. 2004 Sep;66(3):1266-71. doi: 10.1111/j.1523-1755.2004.00881.x. PMID 15327426
- [Background] Movilli E, Gaggia P, Zubani R, Camerini C, Vizzardi V, Parrinello G, Savoldi S, Fischer MS, Londrino F, Cancarini G. Association between high ultrafiltration rates and mortality in uraemic patients on regular haemodialysis. A 5-year prospective observational multicentre study. Nephrol Dial Transplant. 2007 Dec;22(12):3547-52. doi: 10.1093/ndt/gfm466. Epub 2007 Sep 21. PMID 17890254
- [Background] Chamney PW, Kramer M, Rode C, Kleinekofort W, Wizemann V. A new technique for establishing dry weight in hemodialysis patients via whole body bioimpedance. Kidney Int. 2002 Jun;61(6):2250-8. doi: 10.1046/j.1523-1755.2002.00377.x. PMID 12028467
- [Background] Ozkahya M, Ok E, Toz H, Asci G, Duman S, Basci A, Kose T, Dorhout Mees EJ. Long-term survival rates in haemodialysis patients treated with strict volume control. Nephrol Dial Transplant. 2006 Dec;21(12):3506-13. doi: 10.1093/ndt/gfl487. Epub 2006 Sep 25. PMID 17000733
- [Background] Agarwal R, Alborzi P, Satyan S, Light RP. Dry-weight reduction in hypertensive hemodialysis patients (DRIP): a randomized, controlled trial. Hypertension. 2009 Mar;53(3):500-7. doi: 10.1161/HYPERTENSIONAHA.108.125674. Epub 2009 Jan 19. PMID 19153263
- [Background] Charra B. Fluid balance, dry weight, and blood pressure in dialysis. Hemodial Int. 2007 Jan;11(1):21-31. doi: 10.1111/j.1542-4758.2007.00148.x. PMID 17257351
- [Background] Moissl UM, Wabel P, Chamney PW, Bosaeus I, Levin NW, Bosy-Westphal A, Korth O, Muller MJ, Ellegard L, Malmros V, Kaitwatcharachai C, Kuhlmann MK, Zhu F, Fuller NJ. Body fluid volume determination via body composition spectroscopy in health and disease. Physiol Meas. 2006 Sep;27(9):921-33. doi: 10.1088/0967-3334/27/9/012. Epub 2006 Jul 25. PMID 16868355
- [Background] van den Ham EC, Kooman JP, Christiaans MH, Nieman FH, Van Kreel BK, Heidendal GA, Van Hooff JP. Body composition in renal transplant patients: bioimpedance analysis compared to isotope dilution, dual energy X-ray absorptiometry, and anthropometry. J Am Soc Nephrol. 1999 May;10(5):1067-79. doi: 10.1681/ASN.V1051067. PMID 10232694
- [Background] McClanahan BS, Stockton MB, Lanctot JQ, Relyea G, Klesges RC, Slawson DL, Schilling LP. Measurement of body composition in 8-10-year-old African-American girls: a comparison of dual-energy X-ray absorptiometry and foot-to-foot bioimpedance methods. Int J Pediatr Obes. 2009;4(4):389-96. doi: 10.3109/17477160902763358. PMID 19922056
- [Background] Lintsi M, Kaarma H, Kull I. Comparison of hand-to-hand bioimpedance and anthropometry equations versus dual-energy X-ray absorptiometry for the assessment of body fat percentage in 17-18-year-old conscripts. Clin Physiol Funct Imaging. 2004 Mar;24(2):85-90. doi: 10.1111/j.1475-097X.2004.00534.x. PMID 15056180
- [Background] Kraemer M. A new model for the determination of fluid status and body composition from bioimpedance measurements. Physiol Meas. 2006 Sep;27(9):901-19. doi: 10.1088/0967-3334/27/9/011. Epub 2006 Jul 24. PMID 16868354
- [Background] Dou Y, Cheng X, Liu L, Bai X, Wu L, Guo W, Zhao X, Wang F, Cao L, Zuo L. Development and validation of a new dry weight estimation method using single frequency bioimpedance in hemodialysis patients. Blood Purif. 2011;32(4):278-85. doi: 10.1159/000330337. Epub 2011 Aug 26. PMID 21876350
- [Background] Guida B, De Nicola L, Trio R, Pecoraro P, Iodice C, Memoli B. Comparison of vector and conventional bioelectrical impedance analysis in the optimal dry weight prescription in hemodialysis. Am J Nephrol. 2000 Jul-Aug;20(4):311-8. doi: 10.1159/000013606. PMID 10970985
- [Derived] Liu L, Sun Y, Chen Y, Xu J, Yuan P, Shen Y, Lin S, Sun W, Ma Y, Ren J, Liu W, Lei J, Zuo L. The effect of BCM guided dry weight assessment on short-term survival in Chinese hemodialysis patients : Primary results of a randomized trial - BOdy COmposition MOnitor (BOCOMO) study. BMC Nephrol. 2020 Apr 15;21(1):135. doi: 10.1186/s12882-020-01793-x. PMID 32295531
- [Derived] Liu L, Long G, Ren J, Li J, Xu J, Lei J, Li M, Qiu M, Yuan P, Sun W, Lin S, Liu W, Sun Y, Ma Y, Mao Y, Shen Y, Zuo L. A randomized controlled trial of long term effect of BCM guided fluid management in MHD patients (BOCOMO study): rationales and study design. BMC Nephrol. 2012 Sep 25;13:120. doi: 10.1186/1471-2369-13-120. PMID 23006960